CLINICAL TRIAL: NCT03540927
Title: Impact of a Multicomponent Group Intervention on Psychosocial Well-being of Rehabilitated Entrepreneurs in a Conflict-affected Area of Pakistan: A Randomised Controlled Trial
Brief Title: Problem Management Plus for Entrepreneurs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: World Bank (Other); University of Liverpool (Other); Khyber Medical University Peshawar (Other); Institute of Psychitry,WHO Collaborating Centre, Rawalpindi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-WB PM+
Record Dates: First submitted 2018-04-14; First posted 2018-05-30 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Well-being; Psychological Capital; Anxiety; Depression
Keywords: Well-being; Entrepreneurs; Conflict affected settings; Psychosocial intervention; Psychological Capital
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only outcome assessors will be blind to allocation status of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PM+ for entrepreneurs (Experimental): The intervention arm participants will receive a cash transfer to support them in their businesses PLUS 5 weekly face-to-face group sessions of Problem Management Plus(PM+ for entrepreneurs). Duration of each session is 2 hours. Session 1 orients participants to the intervention with motivational interviewing techniques to improve engagement, provides information about common reactions to adversity, and trains participants in a basic stress management strategy (slow breathing). Session 2 discusses problem solving technique.Sessions 3 and 4 support participants' continued application of problem solving, behavioral activation, and stress management and introduce strategies to strengthen social support networks. In session 5, education about retaining intervention gains and self-care are provided and all learned strategies are reviewed.
  Interventions: Behavioral: PM+ for entrepreneurs; Other: Cash transfer to the Entrepreneurs
- Control (Active Comparator): The control arm will receive a cash transfer only to support them in their businesses.
  Interventions: Other: Cash transfer to the Entrepreneurs

INTERVENTIONS:
Behavioral: PM+ for entrepreneurs — The intervention arm will receive 5 weekly face-to-face group sessions of Problem Management Plus(PM+ for entrepreneurs). Duration of each session is 2 hours. Session 1 orients participants to the intervention with motivational interviewing techniques to improve engagement,provides information about common reactions to adversity, and trains participants in a basic stress management strategy (slow breathing). Session 2 addresses a participant-selected problem using problem-solving techniques. Sessions 3 and 4 support participants' continued application of problem solving, behavioral activation, and stress management and introduce strategies to strengthen social support networks. In session 5, education about retaining intervention gains and self-care are provided and all learned strategies are reviewed.
  Arms: PM+ for entrepreneurs
Other: Cash transfer to the Entrepreneurs — The entrepreneurs in the control arm will receive cash transfer only for their businesses.

SUMMARY:
Conflict and unrest over three decades has resulted in significant economic decline in Khyber Pakhtunkhwa (KP) and Federally Administered Tribal Areas (FATA) of Pakistan and these now rank among the poorest regions in the country. The 2009-10 insurgency and subsequent security operations affected both regions and displaced an estimated 2 million people. The severe damage to infrastructure and livelihoods negatively impacted the social and economic fabric of the entire region. As peace has returned to the area, the Economic Revitalization of KP and FATA (ERKF) project, established in 2012 and supported by the World Bank, is working for the rehabilitation of small and medium enterprises (SMEs), with the aim of creation and restoration of jobs. This support is in the form of grants given to individuals who use the funds to establish and run a business in their locality.

Epidemiological studies from the area have shown high rates of common mental disorder (eg., depression, anxiety) in the general population (Husain et al, 2006, Khan et al 2016). Such conditions have a serious impact on the well-being, functioning and productivity of affected individuals (World Health Organization, 2000). For example, in the USA, Depressive Disorders have been estimated to cost the economy over US$210 billion per annum, largely due to reduced productivity (Greenberg et al, 2015). The economic rehabilitation of a population exposed to a humanitarian crisis, and therefore at greater risk of depression, must include interventions to reduce mental morbidity so the individuals are able to function better and potentially improve their long-term productivity.

The Human Development Research Foundation, in collaboration with the World Bank, has adapted a 5-session group intervention from WHO Problem Management Plus program, tailored to the needs of small and medium enterprise owners affected by the prolonged conflict in KP and FATA areas of Pakistan. This intervention (Problem Management Plus adapted for entrepreneurs) is based on established cognitive behavioral strategies previously tested in Pakistan (Rahman et al, 2016). The goal of the intervention is to improve psychological capital,reduce psychosocial distress leading to, increased productivity in the long-term. The intervention will be evaluated using a two arm, single blind randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All small and medium entrepreneurs, leading SMEs and family businesses in situations of fragility encountered in KP/FATA, Pakistan, who received a cash transfer for rehabilitation of their businesses by Economic Revitalization of Khyber Pakhtunkhwa and FATA (ERKF), Pakistan.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Primary end point is percentage change in the prevalence of psychological distress in the intervention arm as compared to the control arm at 3 months post intervention.
  The primary outcome is change in the prevalence of psychological distress as measured by PHQ-9 in the intervention arm as compared to the control arm. The 9-item Patient Health Questionnaire (PHQ-9), incorporates DSM-IV depression diagnostic criteria with other key major depressive symptoms (Kroenke et al, 2001). Participants rate their responses on a 4-point Likert scale ranging from not at all to nearly every day. The PHQ-9 total severity score ranges from 0 to 27. The PHQ-9 has been validated in the Urdu language, showing adequate sensitivity and specificity (Husain et al 2006) and has been used in recent studies in KP (Rahman et al, 2016).

SECONDARY OUTCOMES:
WHO-5 Well being index (WHO-5) | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  Well-being will be measured by WHO 5 Well-being index (Topp, et al, 2015). WHO-5 is a short and generic global rating scale measuring subjective well-being, the respondent is asked to rate how well each of the 5 statements applies to him or her when considering the last 14 days. The instrument will be administered to study participants at 3 months post intervention to rate their subjective well being in last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). The raw score ranges from 0 (absence of well-being) to 25 (maximal well-being). Scores are then converted to a percentage scale from 0 (absent) to 100 (maximal).
GAD-7 | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  GAD-7 will be used to measure anxiety (Spitzer et al, 2006) in the study sample. GAD-7 is based on the Diagnostic and Statistical Manual of Mental Disorders Version IV (DSM IV) diagnostic criteria for generalised anxiety disorder, and has 7 items. Each item is scored on a likert scale from 0 to 3, generating a maximum score of 21
Psychological Capital Questionnaire | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  Psychological capital will be measured using the Psychological Capital Questionnaire (PCQ) 12 items version (Avey et al, 2007). The PCQ-12 measures psychological capital across four domains (hope-4 items, optimism-2 items, resilience -3 items and self-efficacy-3 items).
Multi-dimensional Scale for Perceived Social Support (MSPSS) | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  Social support will be measured using Multidimensional Scale for Perceived Social Support (MSPSS), adapted for use with this population. MSPSS measure perceived social support in three domains: family, friends and significant others (4 items each). Each item is rated on a seven-point Likert-scale (1 = very strongly disagree; 7 = very strongly agree). A total score is calculated by summing the results for all items (Akhtar et al, 2010; Zimet et al, 1988).
Individual Entrepreneurial Orientation (IEO) | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  Individual entrepreneurial behaviours will be measured using an adapted individual entrepreneurial orientation scale (Lee & Lim, 2009). Data will be collected on autonomy, innovativeness, risk taking, competitive aggressiveness, information seeking (proactive behaviour) and impulsiveness to reflect the degree of change in behaviours
Business behaviors | The secondary outcome data will be collected at 1 week post intervention and at 3 months post intervention
  A specially designed questionnaire will be used to measure behaviours related to business planning.
Long term productivity | 12 months follow-up
  Long-term productivity will be measured using administrative data 12 months post the intervention. This would include data on key business metrics (sales, profits, employee turnover, amount of loans outstanding) as well as whether the firms are innovating or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Development Research Foundation, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan MN, Chiumento A, Dherani M, Bristow K, Sikander S, Rahman A. Psychological distress and its associations with past events in pregnant women affected by armed conflict in Swat, Pakistan: a cross sectional study. Confl Health. 2015 Dec 10;9:37. doi: 10.1186/s13031-015-0063-4. eCollection 2015. PMID 26664447
- [Background] Husain N, Gater R, Tomenson B, Creed F. Comparison of the Personal Health Questionnaire and the Self Reporting Questionnaire in rural Pakistan. J Pak Med Assoc. 2006 Aug;56(8):366-70. PMID 16967789
- [Background] Greenberg PE, Fournier AA, Sisitsky T, Pike CT, Kessler RC. The economic burden of adults with major depressive disorder in the United States (2005 and 2010). J Clin Psychiatry. 2015 Feb;76(2):155-62. doi: 10.4088/JCP.14m09298. PMID 25742202
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Rahman A, Hamdani SU, Awan NR, Bryant RA, Dawson KS, Khan MF, Azeemi MM, Akhtar P, Nazir H, Chiumento A, Sijbrandij M, Wang D, Farooq S, van Ommeren M. Effect of a Multicomponent Behavioral Intervention in Adults Impaired by Psychological Distress in a Conflict-Affected Area of Pakistan: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2609-2617. doi: 10.1001/jama.2016.17165. PMID 27837602
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Akhtar A, Rahman A, Husain M, Chaudhry IB, Duddu V, Husain N. Multidimensional scale of perceived social support: psychometric properties in a South Asian population. J Obstet Gynaecol Res. 2010 Aug;36(4):845-51. doi: 10.1111/j.1447-0756.2010.01204.x. PMID 20666955
- See also: Mental health and work : impact, issues, and good practices — http://www.ilo.org/skills/pubs/WCMS_108152/lang--en/index.htm
- See also: Entrepreneurial orientation and the performance of service business — http://link.springer.com/article/10.1007/s11628-008-0051-5